CLINICAL TRIAL: NCT00995748
Title: REgistry on Cardiac Rhythm disORDers in Asia-Pacific
Brief Title: The RECORD Asia-Pacific Atrial Fibrillation Registry
Acronym: RECORDAF-AP
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: DIREG_R_04434
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Primary objective of this registry is to assess the control of Atrial Fibrillation (AF) over one year in patients attending clinical or specialized practices.

The Secondary objectives are:

* To describe key demographics and treatment features in AF patients visiting cardiologists in various countries in Asia-Pacific.
* To establish correlation between control of AF and clinical outcomes.
* To establish correlation between treatment strategies and AF control.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with either:

  * History of atrial fibrillation diagnosed < 1 year by standard Electro-Cardiogram (ECG) or by ECG-Holter monitoring (treated or not or whatever rhythm at inclusion).
  * New atrial fibrillation diagnosed by standard ECG or by ECG-Holter monitoring at inclusion visit.
* Patient eligible for a pharmacological treatment of AF (by rhythm or rate control agent).

Exclusion Criteria:

* AF due to transient cause (thyrotoxicosis, alcohol intoxication, acute phase of myocardial infarction, pericarditis, myocarditis, electrocution, pulmonary embolism or other pulmonary disease, hydroelectrolytic disorder, metabolic disorder, etc.).
* Post cardiac surgery AF (≤3 months).
* Mentally disabled patients unable to understand or sign the written informed consent.
* Patients unable to comply with follow-up visits.
* Patients with pacemaker, Implantable Cardioverter Defibrillator (ICD).
* Patients scheduled for pulmonary vein ablation, AV node/His bundle ablation, or pacemaker implantation.
* Patient included in any clinical trial in the previous 3 months.
* Pregnant or breastfeeding women.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from office or hospital-based cardiologists from Asia-Pacific countries
Sampling Method: Non-Probability Sample
Enrollment: 2674 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of therapeutic success by patients in sinus rhythm or heart rate control at target (< 80 beats per minute at rest) | At 12 ± 3 months follow-up
Comparison of clinical outcomes (Cardiovascular death, Stroke, Myocardial infarction, etc) for patients in rhythm versus rate control strategies | At 12 ± 3 months follow-up

SECONDARY OUTCOMES:
Treatment effectiveness evaluated by the proportion of patients in sinus rhythm | At 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand